CLINICAL TRIAL: NCT00727324
Title: A Pilot, Open-label, Multi-center Clinical Trial to Investigate the Safety and Efficacy of Bovine-Calf Intestinal Alkaline Phosphatase in Patients With Moderate to Severe Ulcerative Colitis.
Brief Title: Safety/Efficacy Study of Bovine Intestinal Alkaline Phosphatase in Patients With Moderate to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AM-Pharma (Industry)
Collaborators: CRM Biometrics GmbH (Industry); Sintesi Research Srl (Industry); Vigilex BV (Unknown)
Responsible Party: J. Arend, MD, AM-Pharma BV
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AP IBD 02-02
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; UC; moderate; severe; LPS; Alkaline Phosphatase; AP; BIAP; Mucositis
MeSH Terms: conditions — Colitis, Ulcerative; Lymphoma, Follicular; Mucositis | interventions — 2-(3',4'-dihydroxyphenyl-1-azo)benzimidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): BIAP
  Interventions: Drug: bovine intestinal alkaline phosphatase (BIAP)

INTERVENTIONS:
Drug: bovine intestinal alkaline phosphatase (BIAP) — 30,000U/24h for 7 consecutive days via a duodenal catheter
  Other Names: BIAP; AP

SUMMARY:
Ulcerative colitis is characterized by abnormal activation of, and damage to, the colon epithelium, which is considered to be a central pathogenic mechanism. Activation of colon epithelium cells in UC is associated with an abnormal high expression of Toll-like receptors, including TLR-4, the major transducer of LPS, binding specifically the lipid A portion of LPS. Alkaline Phosphatase binds and subsequently dephosphorylates LPS, thereby eliminating the ability of LPS to activate TLR-4. This is expected to 1) prevent activation of the intestinal epithelium and 2) prevent systemic inflammatory responses that result from transmigration of endotoxin though the leaky inflamed intestinal mucosa. Therefore, it is expected that administration of BIAP may attenuate or prevent the local and systemic inflammatory response in patients with severe ulcerative colitis.

DETAILED DESCRIPTION:
Inflammatory Bowel Disease (IBD) is a general term for a group of non-specific, chronic inflammatory disorders of the digestive tract, of unknown etiology. IBD may be divided in two major categories: Ulcerative colitis and Crohn's disease, both characterized by a tendency towards frequent acute relapses leading to devastating chronic destruction of the intestinal mucosal barrier function. Whereas Crohn's disease can affect the whole digestive tract, ulcerative colitis is characterized by colonic involvement only. Surgical intervention is frequently required in both Crohn's disease and ulcerative colitis. Therapeutic intervention to date predominantly is based on reduction of induced local mucosal- or systemic inflammation by the use of 5-ASA, corticosteroids, cyclosporine, or TNFα antibodies.

In IBD, the delicate balance between pro-inflammatory molecules, anti-inflammatory molecules and immunoregulatory cells, which tightly regulate the immune system, is disrupted and this results in chronic, relapsing inflammation. Tissue and plasma concentrations of pro-inflammatory cytokines such as IFN-gamma, IL-1ß, IL-6, IL-8 and TNFα are elevated in inflammatory bowel disease and correlate with IBD activity.

In patients with inflammatory bowel diseases circulating LPS have been detected and also increased AP levels have been observed. The presence of the endotoxin is probably the consequence of the damaged intestinal mucosa leading to an increased LPS influx or gut translocation and causing or aggravating the systemic inflammatory response. The increased AP levels observed in these patients may be caused by the suboptimal detoxification of the gut-derived influx of LPS and a response thereof of non-intestinal organs. Thus it has been proposed that the liver sheds alkaline phosphatase (fast acting liver alkaline phosphatase) massively after having been insulted with LPS.

Systemic consequences of IBD may be induced and/or aggravated significantly by the influx of LPS. The proposed normal natural defense mechanism against LPS does include, amongst others, the cleavage of one of the phosphate groups from LPS by endogenous AP. It is therefore conceivable that a reduction in the amount of active LPS in the intestinal lumen by exogenously administered AP will result in a corresponding relative decrease of LPS-influx in the circulation of a subject and, as a consequence, inhibit the LPS medicated systemic inflammatory response. Moreover, dephosphorylated LPS will reduce the ability of LPS to activate TLR-4, resulting in decreased nuclear factor κB activation and a decreased local inflammatory response.

In order to investigate the clinical potential of exogenously administered BIAP for human use, its safety, tolerability and pharmacokinetics have previously been studied in animal toxicology studies and in subsequent Phase I and IIa clinical trials, respectively. These studies were done with intravenously administered BIAP. Following these studies and the successful completion of animal pharmacology studies and a human volunteer study with oral AP the next phase in the development of exogenously administered oral AP is to test the compound in a limited population of patients with IBD.

ELIGIBILITY:
Inclusion Criteria:

* Age, >18 years, AND
* Capable of understanding the purpose and risks of the study and have provided a signed and dated written IC, AND
* Prior to the study baseline, been treated with oral steroid medication, of which > 2 weeks on oral prednisone equivalent of at least 40mg/day, and still have:

  * active ulcerative colon disease documented by a MAYO score of 6-11, and
  * active ulcerative colon disease documented by a MTWSI score of 7-15

OR

* Prior to the study baseline, documented clinical inability to decrease or stop the course of oral steroid medication. Subjects have been treated for a minimum of 12 weeks, and still have:

  * chronic active ulcerative colon disease documented by a MAYO score of 6-11, and
  * chronic active ulcerative colon disease documented by a MTWSI score of 7-15

OR

* Prior to the study baseline, been treated with a stable dosage of azathioprine for a minimum of 12 weeks, and have a moderate to severe relapse defined as:

  * chronic active ulcerative colon disease documented by a MAYO score of 6-11, and
  * chronic active ulcerative colon disease documented by a MTWSI score of 7-15.

Exclusion Criteria:

* UC, requiring immediate surgical, endoscopic, or radiological intervention; including massive haemorrhage, perforation and sepsis, suppurative complications (intra-abdominal or peri-anal abscesses) or toxic colon,
* history of large bowel surgery,
* history of serious infections,
* positive stool cultures, including Clostridium difficile,
* significant organ dysfunction,
* pregnancy, nursing mothers, or women of childbearing potential without appropriate use of contraceptives,
* treatment with:

  1. an altered dose of any 5-ASA preparation within 4 weeks of screening,
  2. an altered dose of azathioprine or mercaptopurine within 4 weeks of screening (stable dosage of immunosuppressives is allowed), or start of azathioprine in the last 3 months prior to baseline,
  3. probiotics, antibiotics within 1 month, methotrexate or cyclosporine within 2 months prior to screening,
  4. any experimental treatment for this population e.g. infliximab, tacrolimus, FK506 or other anti TNFα therapy) within 2 months of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-05; Primary Completion 2006-11 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Investigate the safety and tolerability of 7 days of BIAP administration in subjects with moderate to severe ulcerative colitis | 28 days

SECONDARY OUTCOMES:
To evaluate the efficacy of 7 days of BIAP administration in subjects with moderate to severe ulcerative colitis | 63 days (9 weeks)
To evaluate the efficacy of 7 days of BIAP administration on related variables in subjects with moderate to severe ulcerative colitis | 63 days (9 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Prof Milan Lukas, PhD, MD, Principal Investigator — University Prague, Czech Republic; Prof Paolo Gionchetti, PhD, MD, Principal Investigator — Policlinico S. Orsola, Bologna, Italy
Locations (11):
- Czechia (4):
  - Internal Clinic, Vitkovice Hospital Ostrava, Ostrava, Vitkovice
  - Teaching Hospital Olomouc, Dep. Internal Clinic, Olomouc
  - Center of Gastroenterology at General Teaching Hospital, Prague
  - Institute of Clinical and Preventive Medicine (IKEM), Clinic of Hepatogastroenterology, Prague
- Italy (7):
  - Università di Ancona - Nuovo Complesso Didattico, Facoltà di Medicina e Chirurgia, Clinica di Gastroenterologia, Ancona, Torrette
  - University of Bologna, Dept of Internal Medicine and Gastroenterology, Bologna
  - Ospedale di Marsciano, Ambulatorio Gastroenterologia, Marsciano
  - Ospedale Santa Maria delle Croci, Servizio di Gastroenterologia e Endoscopia Digestiva, Ravenna
  - Università Cattolica di Roma, Dipartimento di Medicina Interna, Roma
  - Azienda Ospedaliera S. Camillo - Forlanini, Roma
  - Ospedale Mauriziano, UOA Gastroenterologia, Torino

REFERENCES:
- [Background] Poelstra K, Bakker WW, Klok PA, Kamps JA, Hardonk MJ, Meijer DK. Dephosphorylation of endotoxin by alkaline phosphatase in vivo. Am J Pathol. 1997 Oct;151(4):1163-9. PMID 9327750
- [Background] Nakamura M, Saito H, Kasanuki J, Tamura Y, Yoshida S. Cytokine production in patients with inflammatory bowel disease. Gut. 1992 Jul;33(7):933-7. doi: 10.1136/gut.33.7.933. PMID 1644332
- [Background] Brynskov J, Nielsen OH, Ahnfelt-Ronne I, Bendtzen K. Cytokines (immunoinflammatory hormones) and their natural regulation in inflammatory bowel disease (Crohn's disease and ulcerative colitis): a review. Dig Dis. 1994 Sep-Oct;12(5):290-304. doi: 10.1159/000171464. PMID 7882549
- [Result] Lukas M, Drastich P, Konecny M, Gionchetti P, Urban O, Cantoni F, Bortlik M, Duricova D, Bulitta M. Exogenous alkaline phosphatase for the treatment of patients with moderate to severe ulcerative colitis. Inflamm Bowel Dis. 2010 Jul;16(7):1180-6. doi: 10.1002/ibd.21161. PMID 19885903
- See also: AM-Pharma Homepage — http://www.am-pharma.com